CLINICAL TRIAL: NCT05930470
Title: Pilot-testing the Effect of Magnetic Mitohormesis Therapy for Treating Frailty in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Auburn University (Other)
Collaborators: QuantumTX Pte Ltd (Network)
Responsible Party: Principal Investigator, Andrew Fruge, Assistant Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AU MMT 23
Record Dates: First submitted 2023-04-19; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Frailty
Keywords: frailty; aging; physical performance
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Sham-controlled crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed intervention (Sham Comparator): Sham treatment first, then Magnetic Mitohormesis Therapy treatment
  Interventions: Other: Magnetic Mitohormesis Therapy
- Immediate intervention (Experimental): Magnetic Mitohormesis Therapy treatment first, then Sham treatment
  Interventions: Other: Magnetic Mitohormesis Therapy

INTERVENTIONS:
Other: Magnetic Mitohormesis Therapy — The MMT device that will be used in the trial will be the QuantumTx BIXEPS Fitness and Wellness. The apparatus will provide pulsed electromagnetic fields at flux densities 1.5 mT. During the treatment period, participants will receive PEMF therapy during two ten-minute sessions each week for a total of 12 weeks. The treatment period will be preceded or followed by 12 weeks of twice-weekly sham treatments depending on randomization.
  Other Names: Pulsed Electromagnetic Field Therapy

SUMMARY:
Thirty (30) adults with limited physical function will be recruited to participate in a double-blind pilot randomized controlled crossover trial in which all participants will receive 12-weeks of twice weekly MMT treatment in the first (Phase 1) or second half (Phase 2) of the study period; during the control period, participants will receive sham treatment and will be blinded to the randomization.

ELIGIBILITY:
Inclusion Criteria:

* physical frailty or pre-frailty, indicated by Short Physical Performance Battery Score <10;
* intact cognition indicated by a Mini-Cog Screening Test Score > 2;
* able to read and write in English; and
* access to a telephone.

Exclusion Criteria:

* active malignancy;
* neuro-degenerative disease
* active electronic implants;
* any health conditions that would prevent performing the testing and intervention procedures;
* major surgical procedures within the last 6 months;
* major change in prescription medications within the last 3 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of adherence to intervention | 24 weeks
  75% session attendance
Number of sites successfully recruited | 1 year
  Study recruitment, intervention, and data collection will be conducted at independent and assisted living facilities. Thus, reaching target accrual requires successful recruitment of these facilities. This outcome measures the actual number of study sites/facilities agreeing to and providing physical access and support to conduct the study.
Likert scale assessment of protocol implementation | 1 year
  Study staff assessment of device usability and assessment protocol. Two questions with likert scale responses ranging from 1-5, with a higher score meaning a better outcome.
Likert scale assessment of participant satisfaction | 24 weeks
  Participant Satisfaction Survey. Eight questions with likert scale responses ranging from 1-5, with a higher score meaning a better outcome.

SECONDARY OUTCOMES:
Objective Frailty - Short Physical Performance Battery (SPPB) | Change from 0-12 weeks, 12-24 weeks
  Repeated Chair stand, balance test, and 4-meter walk composite score (0-12), with higher scores indicating a better outcome
Physical activity - accelerometry | Change from 0-12 weeks, 12-24 weeks
  Number of daily steps, with higher scores indicating a better outcome
Grip strength | Change from 0-12 weeks, 12-24 weeks
  handheld dynamometry, with higher scores indicating a better outcome
Quality of Life T-score | Change from 0-12 weeks, 12-24 weeks
  Research ANd Development (RAND) Short Form-12 will assess mental and physical quality of life, with higher scores indicating a better outcome
Subjective Frailty score (0-5) | Change from 0-12 weeks, 12-24 weeks
  Frail questionnaire, with higher scores indicating a better outcome
SWAY Memory Score | Change from 0-12 weeks, 12-24 weeks
  SWAY Memory Test Score, ranging from 0-100, with higher scores indicating a better outcome
Body composition | Change from 0-12 weeks, 12-24 weeks
  Body Impedence Analyzer (InBody 720) lean body mass (in kilograms)

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Feng Tsai, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venugobal S, Tai YK, Goh J, Teh S, Wong C, Goh I, Maier AB, Kennedy BK, Franco-Obregon A. Brief, weekly magnetic muscle therapy improves mobility and lean body mass in older adults: a Southeast Asia community case study. Aging (Albany NY). 2023 Mar 19;15(6):1768-1790. doi: 10.18632/aging.204597. Epub 2023 Mar 19. PMID 36934330
- [Background] Stephenson MC, Krishna L, Pannir Selvan RM, Tai YK, Kit Wong CJ, Yin JN, Toh SJ, Torta F, Triebl A, Frohlich J, Beyer C, Li JZ, Tan SS, Wong CK, Chinnasamy D, Pakkiri LS, Lee Drum C, Wenk MR, Totman JJ, Franco-Obregon A. Magnetic field therapy enhances muscle mitochondrial bioenergetics and attenuates systemic ceramide levels following ACL reconstruction: Southeast Asian randomized-controlled pilot trial. J Orthop Translat. 2022 Oct 13;35:99-112. doi: 10.1016/j.jot.2022.09.011. eCollection 2022 Jul. PMID 36262374
- [Background] Yap JLY, Tai YK, Frohlich J, Fong CHH, Yin JN, Foo ZL, Ramanan S, Beyer C, Toh SJ, Casarosa M, Bharathy N, Kala MP, Egli M, Taneja R, Lee CN, Franco-Obregon A. Ambient and supplemental magnetic fields promote myogenesis via a TRPC1-mitochondrial axis: evidence of a magnetic mitohormetic mechanism. FASEB J. 2019 Nov;33(11):12853-12872. doi: 10.1096/fj.201900057R. Epub 2019 Sep 13. PMID 31518158
- [Background] Tai YK, Ng C, Purnamawati K, Yap JLY, Yin JN, Wong C, Patel BK, Soong PL, Pelczar P, Frohlich J, Beyer C, Fong CHH, Ramanan S, Casarosa M, Cerrato CP, Foo ZL, Pannir Selvan RM, Grishina E, Degirmenci U, Toh SJ, Richards PJ, Mirsaidi A, Wuertz-Kozak K, Chong SY, Ferguson SJ, Aguzzi A, Monici M, Sun L, Drum CL, Wang JW, Franco-Obregon A. Magnetic fields modulate metabolism and gut microbiome in correlation with Pgc-1alpha expression: Follow-up to an in vitro magnetic mitohormetic study. FASEB J. 2020 Aug;34(8):11143-11167. doi: 10.1096/fj.201903005RR. Epub 2020 Jul 6. PMID 32627872